CLINICAL TRIAL: NCT03054935
Title: The Effects of Disease Activity on Resting Energy Expenditure in Subjects With Crohn's Disease: A Cross-sectional Study
Brief Title: Resting Energy Expenditure Evaluation in Subjects With Crohn's Disease
Acronym: REECD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fabrizio Pasanisi (Other)
Collaborators: Fabiana Castiglione (Unknown)
Responsible Party: Sponsor-Investigator, Fabrizio Pasanisi, Associate Professor of Internal Medicine, Federico II University
Organization: Federico II University (Other)
Other Study IDs: 102/16
Record Dates: First submitted 2017-02-08; First posted 2017-02-16 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Crohn Disease
Keywords: Energy Expenditure; Body Composition; Food Intake
MeSH Terms: conditions — Crohn Disease | interventions — Calorimetry, Indirect

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subject-CD: Subjects with Crohn's Disease in active or quiescent phase, classified according to Crohn's Disease Activity Index (CDAI >150 active; CDAI < 150 quiescent)
  Interventions: Other: Indirect Calorimetry

INTERVENTIONS:
Other: Indirect Calorimetry — Measurement of resting energy expenditure

SUMMARY:
The aim of this study is to investigate the effect disease activity on resting energy expenditure (REE), body composition, inflammatory markers, food intake and quality of life in subjects affected by Crohn's Disease (CD)

DETAILED DESCRIPTION:
Malnutrition is a common sequel among patients affected by Crohn's disease (CD). The pathogenic mechanisms include poor dietary intake, increased resting energy expenditure (REE), nutrient malabsorption and loss. So far, few studies have been carried out in CD adult patients, assessing the effect of disease activity on both REE and body composition. Vaisman et al (2006) studied sixteen CD patients in remission (> 3 mo) and showed no effect of REE on lower BMI, although in the presence of similar energy intake in according with previous studies (Al-Jaouni et al., 2000; Schneeweiss et al., 1999). While, Gong et al., 2015 found that patients with active disease had an increase in REE compared to patients in remission as already shown by Rigaud et al., 1993; Kushner and Schoeller, 1991. Overall, the effect of disease activity on REE is still uncertain and requires further investigation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Crohn's Disease

Exclusion Criteria:

* Comorbidity affecting energy metabolism (diabetes mellitus, thyroid dysfunction, etc.)
* History of acute or chronic liver or kidney disease
* Current parenteral nutrition
* Presence of fistulae, ileostomy or colostomy
* Presence of extensive small bowel resection (residual small bowel < 2 meters)
* Pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending Gastroenterology Unit
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Resting Energy Expenditure (REE) measured by Indirect Calorimetry (IC) in patients with Crohn's Disease | At baseline
  The measurement of REE by IC is a non-invasive method that measures oxygen consumption and carbon dioxide production and it is generally considered the gold standard in clinical practice.

SECONDARY OUTCOMES:
Body composition assessment by bioelectrical impedence analysis (BIA) | At baseline
Assessment of muscle function by hand-grip strength | At baseline
  Hand-grip strength will be performed by dynamometer
Food intake evaluation | At baseline
  Food intake will be assessed by filling 3 day food records
Inflammatory biomarkers | At baseline
  Serum concentration of high sensitive C-reactive protein (hs-RCP) will be determined by immunoturbidimetric assay while tumor necrosis factor - alpha (TNF-alpha) and Interleukin 6 (IL-6) will be assessed by ELISA.
Quality of Life (QoL) | At baseline
  Assessment of each patient's health and well-being using the short-form 36 (SF-36).

CONTACTS AND LOCATIONS:
Locations (1):
- Federico II University Hospital, Napoli, Italy

REFERENCES:
- [Background] Al-Jaouni R, Hebuterne X, Pouget I, Rampal P. Energy metabolism and substrate oxidation in patients with Crohn's disease. Nutrition. 2000 Mar;16(3):173-8. doi: 10.1016/s0899-9007(99)00281-6. PMID 10705071
- [Background] Gong J, Zuo L, Guo Z, Zhang L, Li Y, Gu L, Zhao J, Cao L, Zhu W, Li N, Li J. Impact of Disease Activity on Resting Energy Expenditure and Body Composition in Adult Crohn's Disease: A Prospective Longitudinal Assessment. JPEN J Parenter Enteral Nutr. 2015 Aug;39(6):713-8. doi: 10.1177/0148607114528360. Epub 2014 Mar 25. PMID 24668997
- [Background] Kushner RF, Schoeller DA. Resting and total energy expenditure in patients with inflammatory bowel disease. Am J Clin Nutr. 1991 Jan;53(1):161-5. doi: 10.1093/ajcn/53.1.161. PMID 1984342
- [Background] Rigaud D, Cerf M, Angel Alberto L, Sobhani I, Carduner MJ, Mignon M. [Increase of resting energy expenditure during flare-ups in Crohn disease]. Gastroenterol Clin Biol. 1993;17(12):932-7. French. PMID 8125226
- [Background] Schneeweiss B, Lochs H, Zauner C, Fischer M, Wyatt J, Maier-Dobersberger T, Schneider B. Energy and substrate metabolism in patients with active Crohn's disease. J Nutr. 1999 Apr;129(4):844-8. doi: 10.1093/jn/129.4.844. PMID 10203559
- [Background] Vaisman N, Dotan I, Halack A, Niv E. Malabsorption is a major contributor to underweight in Crohn's disease patients in remission. Nutrition. 2006 Sep;22(9):855-9. doi: 10.1016/j.nut.2006.05.013. PMID 16928471